CLINICAL TRIAL: NCT00476255
Title: Evaluating Models for Dissemination of Injury Prevention Information in the PED
Brief Title: Evaluating Models for Dissemination of Injury Prevention Information in the Pediatric Emergency Department Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfunded
Sponsor: Rhode Island Hospital (Other)
Responsible Party: James G. Linakis, PhD, MD, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0080-06
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2010-04

CONDITIONS: Car Seats; Injuries
Keywords: child safety restraint; injury prevention; automotive
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Standard Care (Active Comparator): Instructional materials
  Interventions: Behavioral: Enhanced Standard Care (ESC)
- Motivational Intervention (Experimental): Motivational interview
  Interventions: Behavioral: Brief Motivational Intervention (BMI)

INTERVENTIONS:
Behavioral: Enhanced Standard Care (ESC) — Reading material
  Arms: Enhanced Standard Care
Behavioral: Brief Motivational Intervention (BMI) — Motivational interview with trained therapist
  Arms: Motivational Intervention

SUMMARY:
This study examines the Pediatric Emergency Department as a location for increasing safe car seat practices by parents who are not restraining their children appropriately in motor vehicles. Three different intervention will be tested to determine their effectiveness in increasing safe car seat practices: usual emergency department care; provision of printed materials; and a brief motivational intervention in the emergency department.

DETAILED DESCRIPTION:
The long-term goal of the present research program is to enhance the utilization of evidence-based injury prevention strategies and to encourage medical practitioners to disseminate focused information regarding injury prevention in the Pediatric Emergency Department (ED). This study examines the Pediatric Emergency Department as a location for increasing safe car seat practices by parents who are not restraining their children appropriately in motor vehicles. Three different intervention will be tested to determine their effectiveness in increasing safe car seat practices. The proposed research plan: 1. examines the efficacy of a Brief Motivational Intervention to enhance automobile safety restraint-specific injury prevention behaviors in parents/caregivers of younger children; and 2. examines the efficacy of focused, behavior-specific, injury prevention discharge instruction supplements (Enhanced Standard Care) in increasing safety restraint-specific injury prevention behaviors in parents/caregivers of younger children. We will conduct a randomized, controlled trial of parent/caregivers of children being evaluated in the Hasbro Children's Hospital Emergency Department in Providence, Rhode Island. Eligible, consenting participants will be screened with an injury assessment tool for inappropriate use of motor vehicle child safety restraints. High risk participants will be randomized into three intervention groups: Standard Care (SC), Enhanced Standard Care (ESC) and Brief Motivational Intervention (BMI). All participants will then be contacted three months following enrollment and surveyed regarding child safety restraint practices, attitudes and knowledge. The following main effects will be evaluated with relation to child safety restraint practice and attitude change: 1. Intervention (SC vs. ESC vs. BMI); 2. Injury status of child (Injured vs. non-injured). In addition, we will monitor re-injury rates of the index children of all enrolled parent/caregivers for one year from the time of enrollment and compare on the bases of the above main effects.

ELIGIBILITY:
Inclusion Criteria:

* Parents/primary caregivers of children ages 0-7 years who are being seen in the Pediatric ED for a non life-threatening injury or non-injury related complaint
* Parents/primary caregivers whose children are medically stable
* Parent/primary caregiver has legal custody of the index child and is able to provide informed consent for participation
* Parent/primary caregiver speaks English or Spanish
* Parent/primary caregiver must have access to a motor vehicle in which the child is transported

Exclusion Criteria:

* parents/primary caregivers who are cognitively unable to take part in the intervention
* those whose children are suspected by the clinical staff of being victims of child abuse
* those whose children are medically or surgically unstable
* those whose children are being evaluated for possible psychiatric disorders or suicidal ideation
* those who do not speak English or Spanish, and those without a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Self-reported child safety restraint practices, attitudes and knowledge | 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: James G Linakis, PhD, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States